CLINICAL TRIAL: NCT06412458
Title: Phase I Clinical Study to Evaluate the Safety and Efficacy of IM83 CAR-T Cells for the Treatment of Relapsed or Refractory Osteosarcoma
Brief Title: IM83 Clinical Study of CAR-T Cell Therapy in Patients With Relapsed or Refractory Osteosarcoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM83-002
Record Dates: First submitted 2024-04-23; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Refractory Osteosarcoma; Recurrent Osteosarcoma
Keywords: IM83 CAR-T; Relapsed or refractory osteosarcoma
MeSH Terms: conditions — Osteosarcoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM83 CAR-T Cells (Experimental): After preconditioning with chemotherapy, IM83 CAR-T Cells will be evaluated
  Interventions: Biological: IM83 CAR-T Cells

INTERVENTIONS:
Biological: IM83 CAR-T Cells — IM83 CAR-T Cells, 5×10^8 cells, 1×10^9 cells, and 2×10^9 cells, treatment follows a lymphodepletion. Drug: Fludarabine Recommendation: 30 mg/m^2 (D-5~D- 3), determined by tumor burden at baseline. Drug: Fludarabine Recommendation: 30 mg/m^2 (D-5~D-3), determined by tumor burden at baseline. Drug: Cyclophosphamide Recommendation: 300 mg/ m^2 (D-5~D-3), determined by tumor burden at baseline.

SUMMARY:
The purpose of this study, a single-center, open, single-dose clinical study, was to evaluate the safety, tolerability, and pharmacokinetic profile of IM83 CAR-T cells in the treatment of patients with relapsed or refractory osteosarcoma

DETAILED DESCRIPTION:
This study is planned to enroll 9-18 patients with relapsed or refractory osteosarcoma in a modified "3+3" design for dose escalation, with three dose groups of 5×10^8 cells, 1×10^9 cells, and 2×10^9 cells.3-6 subjects are planned to be enrolled in each dose group to assess their safety. Each dose group is planned to enroll 3-6 subjects to assess safety, and if the incidence of horizontal dose-limiting toxicity (DLT) is ≤1/6 within 28 days after transfusion in a dose group, the transfusion of cells from the next dose group can be initiated.

This study will be divided into a screening period, a cell collection period, a chemotherapy pretreatment period, a return infusion and a follow-up period, and within 28 days of return infusion the investigator will assess whether a DLT (Dose limited toxicity) event has occurred to confirm the safety of this dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years, both male and female;
2. Subjects with a diagnosis of osteosarcoma of the extremity confirmed by pathohistologic examination;
3. To enroll subjects with recurrent or refractory extremity osteosarcoma who have failed or are intolerant to first-line standard therapy and who are not candidates for radical surgery and/or localized therapy and who lack effective subsequent treatment.

Notes:

1. Standard treatment failure was defined as disease relapse or progression during or within 6 months of completion of treatment with first-line chemotherapeutic agents (including high-dose methotrexate, doxorubicin, cisplatin, isocyclophosphamide, etc.);
2. Requirement of treatment intolerance: means that the subject is unable to continue the current effective systemic regimen due to the development of toxic side effects such as ≥ grade 3 vomiting, diarrhea, abdominal pain, myelosuppression, etc., and that refusal is not accepted for financial and personal reasons;
3. The standard treatment received by the subject must be in accordance with the Chinese Society of Clinical Oncology (CSCO) Guidelines for the Treatment of Bone and Soft Tissue Tumors, 2023 Edition; 4. At least one measurable target lesion according to RECIST 1.1 criteria; 5. Subjects must provide a tumor tissue sample (paraffin block or number of unstained sections meeting the testing requirements specified by the Institute) within 2 years that meets the requirements to be tested by immunohistochemistry for GPC3 and CD40 and needs to be positive for GPC3 expression;; 6. Karnofsky functional status score ≥60; 7. Expected survival ≥ 12 weeks; 8. Laboratory tests should meet at least the indicators specified below:

1)Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; 2)Absolute lymphocyte cell count (LY) ≥ 0.6 x 10^9/L; 3)Lymphocytes make up ≥10% of white blood cells; 4)Platelets ≥75 x 10^9/L; 5)Hemoglobin ≥ 90 g/L; 6)Creatinine clearance ≥60 ml/min; 7)Serum bilirubin ≤ 1.5 times the upper limit of normal; if liver metastases are present, serum bilirubin ≤ 3.0 times the upper limit of normal; 8)Prolongation of prothrombinogen time ≤ 4s; 9)≤ 2.5 times the upper limit of normal for albumin transaminase (AST) and albumin transaminase (ALT); if liver metastases are present, ALT and/or AST ≤ 5.0 times the upper limit of normal; 9. Left ventricular ejection fraction was >50%; 10. Oxygen saturation >92% in the non-oxygenated state; 11. Women of childbearing potential who had a negative blood pregnancy test prior to the start of the trial and who agreed to use effective contraception for the duration of the trial up to the last follow-up visit; male subjects whose partners were of childbearing potential agreed to use effective contraception for the duration of the trial up to the last follow-up visit; 12. Vascular access is adequate for cell collection, and lines are available for subjects with existing central venous catheters; 13. I or my legal guardian/proxy agree to participate in this trial and sign the informed consent form.

Exclusion Criteria:

1. Presence of brain metastases;
2. Subjects who have previously received or are awaiting an organ transplant;
3. Toxicity due to prior therapy not stabilized or recovered to ≤ grade 1 (except in cases judged by the investigator to be not clinically significant);
4. Autoimmune diseases requiring systemic immunosuppressive therapy, such as systemic lupus erythematosus, rheumatoid arthritis, and ulcerative colitis, within 2 years prior to the start of screening;
5. Use of any of the following medications or treatments during the designated time period prior to cell collection:

   1. Surgical treatment, interventional therapy, radiotherapy, ablation, and other localized treatments for the study disease within 4 weeks prior to cell collection;
   2. Subjects who have had major surgery or significant trauma within 4 weeks prior to cell collection, or who are expected to require major surgery during the study period;
   3. Immunotherapy with anti-PD1, PD-L1, etc. within 4 weeks prior to cell collection;
   4. Therapeutic doses of corticosteroids have been used within 3 days prior to cell collection. However, topical and inhaled steroids are permitted;
6. Other untreated malignant tumors within the previous 5 years or concurrently, except cervical cancer in situ, basal cell carcinoma of the skin, and ductal carcinoma in situ of the breast;
7. Previously treated with targeted GPC3 therapy (can be enrolled if still positive for GPC3 expression upon testing);
8. Those who have previously received other cellular therapy or genetically modified cellular therapy, such as TCR-T therapy, CAR-T therapy, etc;
9. Prior or clinically significant CNS disorders at screening, such as epilepsy, seizures, cerebrovascular disease (ischemia/hemorrhage/infarction), cerebral edema, reversible posterior leukoencephalopathy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disorders, organic brain syndromes, or psychiatric disorders;
10. Presence of chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), and clinically significant pulmonary function test abnormalities;
11. Subjects assessed by the investigator as having a significant amount of plasmapheresis (e.g., pleural effusion, peritoneal effusion, pericardial effusion) that cannot be controlled with treatment;
12. Medication-uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg) or the presence of clinically significant (e.g., active) cardiovascular disease, such as cerebrovascular accident, myocardial infarction, unstable angina pectoris, or severe cardiac arrhythmia that is uncontrolled with medication or that has a potential impact on the study treatment in the 6 months prior to the date of signing of the informed consent;
13. Subjects who are positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and have a peripheral blood HBV-DNA test higher than the lower limit of detection (HBsAg-positive but with a peripheral blood HBV-DNA test lower than the lower limit of detection according to the Guidelines for the Prevention and Treatment of Chronic Hepatitis B, Version 2022, at least at least 4 weeks of antiviral therapy is required prior to the first administration of the investigational drug, and during the course of the study Ongoing antiviral therapy for 6-12 months with monitoring of HBV DNA, HBsAg, and ALT levels every 1-3 months); Hepatitis C virus (HCV) antibody positive and peripheral blood HCV-RNA test above the lower limit of detection; HIV antibody positive; syphilis antibody positive;
14. Active EBV and cytomegalovirus, defined as subjects with IgM antibody-positive or IgM antibody-negative EBV serum but higher-than-normal EBV-DNA; and cytomegalovirus (CMV) serum IgM antibody-positive or IgM antibody-negative cytomegalovirus but higher-than-normal CMV-DNA;
15. Abnormalities of cardiac function include: long QTc syndrome or QTc interval >480 ms; complete left bundle branch block, degree II/III AV block; severe, uncontrolled arrhythmia requiring pharmacologic therapy; history of chronic congestive heart failure with NYHA class ≥3 (refer to Appendix 3) cardiac ejection fraction less than 50% in the 6 months prior to screening; CTCAE ≥3 grade heart valve disease; myocardial infarction, cardiac angioplasty or stenting, unstable angina, history of severe pericardial disease, or other clinically significant cardiac disease within 6 months prior to screening;
16. Subjects requiring anticoagulation therapy;
17. Subjects requiring long-term antiplatelet therapy;
18. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months prior to initiation of screening;
19. Infections (fungal, bacterial, viral, or other) that require intravenous antimicrobial control or are uncontrollable, for simple urinary tract infections, and for bacterial pharyngitis, may be enrolled if the investigator evaluates that they can be controlled by curative treatment;
20. The presence of any factors affecting compliance with the protocol, or the unwillingness or inability of the subject to comply with the procedures required in the study protocol, as judged by the investigator.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Up to 28 days after CAR-T cell infusion
  Incidence of Adverse Events and Abnormal Findings on Clinically Significant Laboratory Tests Associated with IM83 CAR-T Cell Therapy Within 28 Days of Infusion

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Objective remission rate (ORR) after infusion
Disease control rate (DCR) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Post-infusion disease control rate (DCR)
Duration of response (DOR) | At 28 days, 3 months and 6 months after CAR-T cell infusion
  Duration of disease remission (DoR) after infusion
Progress free survival (PFS) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Progress free survival (PFS) after infusion
Overall Survival (OS) | At 28 days, 3 months, 6 months and 12 months after CAR-T cell infusion
  Overall Survival (OS)
AUC (Area Under Curve) 0-D28 | Up to 28 days after CAR-T cell infusion
  AUC 0-D28 of IM83 CAR-T cells in vivo (peripheral blood) after infusion
AUC (Area Under Curve) 0-D90 | Up to 90 days after CAR-T cell infusion
  AUC 0-D90 of IM83 CAR-T cells in vivo (peripheral blood) after infusion
Cmax (Peak Concentration) | Up to 28 days after CAR-T cell infusion
  Peak Concentrationof IM83 CAR-T cells in vivo (peripheral blood) after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No